CLINICAL TRIAL: NCT03810677
Title: Treatment of Varicose Veins With the ELVeS® Radial® 2ring Slim Fiber. Are There Limitations?
Status: Completed | Type: Observational
Sponsor: be Medical (Industry)
Collaborators: Biolitec AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: ELVeS-01
Record Dates: First submitted 2019-01-11; First posted 2019-01-22 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with varicose veins, eligible for EVLA
  Interventions: Device: ELVeS® Radial® 2ring slim fiber

INTERVENTIONS:
Device: ELVeS® Radial® 2ring slim fiber — Device for endovenous laser ablation manufactured by Biolitec AG company (ELVeS system) - diode laser with a wavelength of 1470 nm

SUMMARY:
This study aims to prove that the ELVeS® Radial® 2ring slim fiber is safe and effective in endovenous laser ablation (EVLA) of varicose veins, with a reliable durability by evaluating procedural details/outcomes, clinical success, anatomic success, pain, post-operative adverse events and re-interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. Patient must sign and date the informed consent form prior to treatment.
3. Presence of unilateral or bilateral primary symptomatic varicose veins (CEAP grade ≥ C2).
4. Patient has an insufficient Great Saphenous Vein (GSV), with or without laser ablation of anterior accessory saphenous vein (AASV), posterior accessory saphenous vein (PASV), and/or Small Saphenous Vein (SSV), with venous symptoms (valve incompetence), suitable for endovenous laser ablation (EVLA).
5. Maximum diameter of the to be treated veins is ≤ 14mm.

Exclusion Criteria:

1. Current deep vein thrombosis.
2. Acute superficial thrombosis.
3. Mean diameter of the to be treated veins > 14mm.
4. Tortuous or very superficial veins considered unsuitable for laser treatment.
5. Recurrent varicose veins.
6. Pregnancy.
7. Coagulopathy or bleeding disorders.
8. Contraindications to the use of general or regional anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with varicose veins, eligible for treatment with EndoVenous Laser Ablation (EVLA).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Anatomic success | at 1 month follow-up
  defined as occlusion of the treated veins and lack of reflux objectified with duplex ultrasonography
Anatomic success | at 12 months follow-up
  defined as occlusion of the treated veins and lack of reflux objectified with duplex ultrasonography

SECONDARY OUTCOMES:
Procedural characteristics | at index-procedure
  Details concerning the index-procedure
Pain scoring using the Visual Analog Scale (VAS) | discharge
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he/she experiences. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
Pain scoring using the Visual Analog Scale (VAS) | at 1 week follow-up
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he/she experiences. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
Clinical success, defined as an objective improvement of clinical outcome after treatment, measured with the Venous Clinical Severity Score (VCSS) | at 1 month follow-up
  The VCSS includes 9 hallmarks of venous disease, each scored on a severity scale from 0 to 3.
Clinical success, defined as an objective improvement of clinical outcome after treatment, measured with the Venous Clinical Severity Score (VCSS) | at 12 months follow-up
  The VCSS includes 9 hallmarks of venous disease, each scored on a severity scale from 0 to 3.
Post-operative adverse events | at 1 week follow-up
  numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Post-operative adverse events | at 1 month follow-up
  numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Post-operative adverse events | at 12 months follow-up
  numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Re-interventions | at 1 week follow-up
  including reason for re-intervention and description of treatment
Re-interventions | at 1 month follow-up
  including reason for re-intervention and description of treatment
Re-interventions | at 12 months follow-up
  including reason for re-intervention and description of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Imelda Hospital, Bonheiden, Antwerp
  - Jessa Hospital, Hasselt, Limburg

REFERENCES:
- [Derived] Verbist J, Laeremans V, Gryffroy F, Van den Eynde W, Heerinckx C, Haesen D. Durability and efficacy of the ELVeS(R) Radial(R) 2ring slim fiber for multiple ablations. Phlebology. 2023 Dec;38(10):641-648. doi: 10.1177/02683555231193883. Epub 2023 Aug 6. PMID 37545129